CLINICAL TRIAL: NCT03132012
Title: Skin Health in Young Adults - Preventing Indoor Tanning and Promoting Sun Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1208010685
Record Dates: First submitted 2017-03-20; First posted 2017-04-27 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Skin Neoplasms
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indoor tanning intervention (Experimental): Web-based intervention modules to discourage tanning.
  Interventions: Behavioral: Indoor tanning intervention
- standard of care control (Active Comparator): General information regarding UV protection measures through an online Qualtrics interface. Content will mirror information provided in brochures typically available in a dermatology office or through skin cancer prevention websites.
  Interventions: Behavioral: Standard of care control

INTERVENTIONS:
Behavioral: Indoor tanning intervention — 6 Web-based modules that focus on preventing skin cancer through sun protection and indoor tanning reduction using the Theory of Planned Behavior and Prospect Theory
  Arms: Indoor tanning intervention
Behavioral: Standard of care control — One website with content similar to those available in dermatology offices on skin cancer prevention
  Arms: standard of care control

SUMMARY:
This is a pilot randomized controlled trial of an Internet-based skin cancer prevention intervention as compared to a standard of care control in 80 non-Hispanic white females ages 20-30.

ELIGIBILITY:
Inclusion Criteria:

* Tanned indoors in past 12 months
* Able to communicate well in English
* Reliable Internet access

Exclusion Criteria:

* History of skin cancer (self-report)

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Intention to indoor tan in next year | Baseline
  Indoor tanning intentions are measured on a scale that ranges from 1 (definitely do not intend to indoor tan) to 7 (definitely do intend to indoor tan).
Intention to indoor tan in next year | 12 Weeks First Follow-up
  Indoor tanning intentions are measured on a scale that ranges from 1 (definitely do not intend to indoor tan) to 7 (definitely do intend to indoor tan).
Intention to indoor tan in next year | 24 Weeks Second Follow-up
  Indoor tanning intentions are measured on a scale that ranges from 1 (definitely do not intend to indoor tan) to 7 (definitely do intend to indoor tan).
Number of indoor tanning sessions in the previous 3 months | 12 weeks preceding baseline
  Self-report measure of number of times indoor tanned, reported retrospectively for the preceding 3 months.
Number of indoor tanning sessions in the previous 3 months | baseline to 12 Weeks (First Follow-up)
  Self-report measure of number of times indoor tanned, reported retrospectively for the preceding 3 months.
Number of indoor tanning sessions in the previous 3 months | From 12 Weeks (first Follow-up) to 24 Weeks (Second Follow-up)
  Self-report measure of number of times indoor tanned, reported retrospectively for the preceding 3 months.

SECONDARY OUTCOMES:
Intention to sunbathe outdoors in the next year | Baseline
  Sunbathing intentions are measured on a scale that ranges from 1 (definitely do not intend to indoor tan) to 7 (definitely do intend to indoor tan).
Intention to sunbathe outdoors in the next year | 12 weeks First Follow-up
  Sunbathing intentions are measured on a scale that ranges from 1 (definitely do not intend to indoor tan) to 7 (definitely do intend to indoor tan).
Intention to sunbathe outdoors in the next year | 24 weeks Second Follow-up
  Sunbathing intentions are measured on a scale that ranges from 1 (definitely do not intend to indoor tan) to 7 (definitely do intend to indoor tan).
Number of outdoor sunbathing sessions in the previous 3 months | 12 weeks preceding baseline
  Self-report measure of number of times sunbathed, reported retrospectively for the preceding 3 months.
Number of outdoor sunbathing sessions in the previous 3 months | baseline to 12 Weeks (First Follow-up)
  Self-report measure of number of times sunbathed, reported retrospectively for the preceding 3 months.
Number of outdoor sunbathing sessions in the previous 3 months | From 12 Weeks (first Follow-up) to 24 Weeks (Second Follow-up)
  Self-report measure of number of times sunbathed, reported retrospectively for the preceding 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale School of Public Health, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided